CLINICAL TRIAL: NCT05565274
Title: Outcome of Combined Tramadol and Paracetamol Versus Pentazocine as Labour Analgesia Among Parturients in the Federal Medical Center, Yenagoa, Bayelsa State, Southern Nigeria: A Randomized Controlled Trial
Brief Title: Outcome of Combined Tramadol and Paracetamol Versus Pentazocine as Labour Analgesia Among Parturients
Acronym: OCTAPPENALA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal Medical Centre, Yenagoa (Other Government)
Responsible Party: Principal Investigator, Andrew Orhorho, Principal Investigator, Federal Medical Centre, Yenagoa
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: FMCY/O&G/OCTAPPENALA/2022
Record Dates: First submitted 2022-09-26; First posted 2022-10-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Labor Pain
Keywords: Tramadol; Paracetamol; Pentazocine; Labour; Analgesia; Efficacy; Safety
MeSH Terms: conditions — Labor Pain; Agnosia | interventions — Pentazocine

STUDY DESIGN:
Intervention Model Description: "Randomized"
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The hospital Pharmacist will prepare the drugs in both arms where the first arm will be 2 ml of 100mg tramadol in 5 ml syringe and 2ml of 600mg Paracetamol in 5 ml syringe as well. The second arm will be 2ml of 30mg pentazocine in 5ml syringe plus 2ml of water for injection. Both arms of the medications will be pre-packed in opaque envelopes and labelled by the pharmacist as either A or B who will take no further part in the study. These will be assigned based on the randomized outcome. The randomization list will be on the possession of research assistant who will take no further part in the study after randomly assigning participants to the study arms till the end of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tramadol plus Paracetamol (Experimental): 2ml of 100mg of intramuscular tramadol plus 2ml of 600mg of intramuscular paracetamol unlabeled
  Interventions: Drug: Pentazocine plus placebo
- Pentazocine plus placebo (Active Comparator): 2ml of 30mg of pentazocine plus 2 ml of water for injection will be administered intramuscularly during labour
  Interventions: Drug: Pentazocine plus placebo

INTERVENTIONS:
Drug: Pentazocine plus placebo — 30mg of pentazocine and 2milliLitre of injection water

SUMMARY:
Labour is a very painful experience and epidural analgesia is considered the gold standard for pain relief in labour. Epidural scarcity, cost and shortage of skilled personnel to administer it is a limitation to it's usage in developing countries. Parenteral opioid analgesics such as pethidine and pentazocine are effective labour analgesia commonly used in developing countries but are limited by their side effects. This limitation in their use call for the need for alternative analgesic with similar or superior analgesic effect but with minimal side effects.The study is aimed at evaluating the efficacy and safety of combined tramadol and paracetamol in reducing labour pain among parturients.

DETAILED DESCRIPTION:
There is paucity of data in our environment looking at the efficacy and safety of combined tramadol and paracetamol in relieving labour pain. This study will offer us great opportunity to evaluate their synergistic effect in labour when compared to the commonly used single opioids such as pethidine or pentazocine.

It would be a double blinded randomized controlled trial. One hundred and sixty-six pregnant eligible women in labour would participate in this study. Participants will be randomized equally into two study arms ( Tramadol plus Paracetamol study arm and Pentazocine study arm) after informed consent. The Tramadol plus Paracetamol study arm will receive 100mg of tramadol plus 600mg of paracetamol intramuscularly in a 2ml and 5ml syringe respectively while the pentazocine study arm will receive 30mg of Pentazocine and 2 milliliters of water for injection as placebo intramuscularly in a 2l and 5 ml syringes respectively. Both drugs will be administered to the participants at 4-6cm cervical dilatation during labour. The outcome measures will be evaluated within 5 hours in labour and an hour immediately after delivery. The need for additional rescue analgesia will be assessed as well. Fetal outcome on both arms will be noted too.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women who presented in spontaneous labour at term, carrying Singleton Live Fetus in Active Phase of Labour with Cervical dilatation of 4-6cm who gave consent to participate in the study

Exclusion Criteria:

* Women with severe medical conditions such as diabetes mellitus, severe pre-eclampsia, cardiac, liver and renal disease
* Preterm Labour
* Intrauterine Fetal Death
* Fetal presentation other than cephalic
* Patients with previous caeserean section
* History of hypersensitivity to paracetamol, tramadol and pentazocine
* Complications such as antepartum haemarrhage, polyhydramnious, premature rupture of membrane
* Use of any kind of analgesia before recruitment
* Multiple gestation
* All other delivery except spontaneous vertex delivery Labour that was induced or augmented

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — All pregnant women who presented in spontaneous labour at term, carrying Singleton Live Fetus in Active Phase of Labour with Cervical dilatation of 4-6cm who gave consent to participate in the study
Enrollment: 166 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
To Evaluate the Number of Participants with Pain After 1 hour of Analgesia Administration | 1 hour post analgesia administration
  Pain was Assessed during Labour 1 hour Post Analgesia Administration using the Numerical Rating Scale for Pain. The Numerical Rating Scale has a minimum score of 0, a maximum score of 10 and a range of 0-10, where higher score means a worse outcome (0=No Pain at all, 5 means Moderate Pain and 10= Worse pain imaginable)
To Evaluate the Number of Participants with Pain After 2 hours of Analgesia Administration | 2 hours post analgesia administration
  Pain was Assessed during Labour 2 hours Post Analgesia Administration using the Numerical Rating Scale for Pain. The Numerical Rating Scale has a minimum score of 0, a maximum score of 10 and a range of 0-10, where higher score means a worse outcome (0=No Pain at all, 5 means Moderate Pain and 10= Worse pain imaginable)
To Evaluate the Number of Participants with Pain After 3 hours of Analgesia Administration | 3 hours post analgesia administration
  Pain was Assessed during Labour 3 hours Post Analgesia Administration using the Numerical Rating Scale for Pain. The Numerical Rating Scale has a minimum score of 0, a maximum score of 10 and a range of 0-10, where higher score means a worse outcome (0=No Pain at all, 5 means Moderate Pain and 10= Worse pain imaginable)
To Evaluate the Number of Participants with Pain 4 hours After Analgesia Administration | 4 hours post analgesia administration
  Pain was Assessed during Labour 4 hours Post Analgesia Administration using the Numerical Rating Scale for Pain. The Numerical Rating Scale has a minimum score of 0, a maximum score of 10 and a range of 0-10, where higher score means a worse outcome (0=No Pain at all, 5 means Moderate Pain and 10= Worse pain imaginable)
To Evaluate the Number of Participants with Pain 5 hours After Analgesia Administration | 5 hours post analgesia administration
  Pain was Assessed during Labour 5 hours Post Analgesia Administration using the Numerical Rating Scale for Pain. The Numerical Rating Scale has a minimum score of 0, a maximum score of 10 and a range of 0-10, where higher score means a worse outcome (0=No Pain at all, 5 means Moderate Pain and 10= Worse pain imaginable)
Number of Participants with Treatment Related Adverse Events on both arms | Time of first analgesia administration to 2 hours Post Delivery
  Number of Participants with Treatment Related Adverse Events such as Nausea, Vomiting, Hypersensitivity Reaction, respiratory depression and any other Adverse Effects from the time of first administation to 2 hours post delivery

SECONDARY OUTCOMES:
Participants with Good Service Satisfaction | First 5 hours Post Delivery
  Good Service Satisfaction among participants was Assessed on both arms of the study using the 5-Point Likert's Scale administered in the first 5 hours of delivery. The 5-Point Likert's Scale contains 5 response Options that consist of two extreme sides and a neutral option at the middle. The 5 responses are; very dissatisfied, Dissatisfied, Neither Dissatisfied or Satisfied, Satisfied and Very Satisfied. Participants responsibility is to choose from any of these responses in the administered questionnaire.
Analgesia Administration to Delivery interval | First 2 hours Post Delivery
  To compare the interval between analgesia administration and the time it took participants to deliver on both arms of the study. This was recorded within the first 2 hours of delivery.
Apgar Scores of the Neonates | At first and fifth minutes after birth
  To Evaluate the well being of Neonates delivered on both arms of the study using the Apgar Scores taken at the first and fifth minutes. Apgar Score has a minimum of 0, a maximum score of 10 and a range of 0-10, where higher score mean a better outcome (0-3= low Apgar Score, 4-6= Moderately Abnormal Apgar Score and 7-10= Good Apgar Score
Special Care Baby Unit Admissions | First 2 hours Post Delivery
  To Evaluate the number of Neonates that were admitted into the Special Care Baby Unit within 2 hours of birth. The Special Care Baby Unit is an intensive care unit where optimal emergency treatment is given to the newborn with health related challenges to increase their chance of survival.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Orhorho, Principal Investigator — Federal Medical Center, Yenagoa Bayelsa State Southern Nigeria

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available by December 2023